CLINICAL TRIAL: NCT06016582
Title: Use of Virtual Reality Medical Hypnosis for Anxiolytic Purposes During Frozen Embryo Transfer - Hypno-TEC Feasibility Study
Brief Title: Use of Virtual Reality Medical Hypnosis for Anxiolytic Purposes During Frozen Embryo Transfer
Acronym: Hypno-TEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0510
Record Dates: First submitted 2023-08-21; First posted 2023-08-29 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Anxiety
Keywords: Virtual Reality Hypnosis; Medical Device; Anxiety; Frozen embryo transfer; Feasibility
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients benefiting from the virtual reality hypnosis headset during frozen embryo transfer (Other): The study will involve women, aged between 18 and 45, receiving care within the Reproductive Medicine Department at the Mother-Child-Woman Hospital in Lyon, as part of an assisted reproduction journey, and for whom a frozen embryo transfer is planned. The patients should have previously undergone an embryo transfer to be familiar with the medical procedure to be performed. Their partner must have planned to be present during the FET, in order to comply to identity vigilance regulations.
  The study will be proposed to them during the consultation scheduled for the dispensing of their prescriptions in preparation for the transfer. If the patient agrees to participate, she will then use a virtual reality hypnosis headset during her frozen embryo transfer.
  Interventions: Device: Use of virtual reality hypnosis headset during frozen embryo transfer

INTERVENTIONS:
Device: Use of virtual reality hypnosis headset during frozen embryo transfer — The virtual reality hypnosis headset will be used before, during, and after the FET procedure:
  * The headset will be put on 5 minutes prior to the procedure, allowing time for immersion in the virtual world.
  * The headset will be kept on throughout the entire procedure (procedure duration less than 5 minutes).
  * The headset will be worn for up to 5 minutes after the procedure. The patient will be free to choose her own auditory and visual scenario for the session.
  Prior to the procedure and the device setup, the patient will be asked to complete a self-assessment anxiety questionnaire, the State-Trait Anxiety Inventory. This self-assessment questionnaire is a validated and standardized tool designed to measure temporary "state" anxiety related to a specific situation (in this case, the embryo transfer). After the procedure, the patient will need to complete the questionnaire again, along with another set of questions specifically designed for our study.

SUMMARY:
Assisted Reproduction Technology (ART) procedures are often long and particularly stressful for couples. The level of anxiety appears to persist throughout the entire process, particularly during embryo transfer, a pivotal and delicate stage in In Vitro Fertilization (IVF). Many women apprehend this maneuver, firstly, as it represents the culmination of the process and consequently elicits apprehensions regarding negative outcome, and secondly, as it instigates anxiety related to potential discomfort during the procedure.

Medical Hypnosis in Virtual Reality is a combination of hypnotherapy and immersion in a fictitious world, used in the medical field for anxiolytic and analgesic purposes. This fusion is made possible by a virtual reality headset coupled with an auditory device.

The diversion and relaxation conferred by this device can lead to a reduction in perceived anxiety and an indirect enhancement of compliance and cooperation during medical procedure. Several studies have already demonstrated a benefit on pre-operative and peri-operative anxiety, with reassuring safety data on the use of this medical device.

However, despite the common use of VRH in the medical field, encouraging data on anxiety reduction, and accessibility to these headsets within in certain ART departments, they are not routinely employed during embryo transfers. Various barriers to the implementation of this medical device in this indication seem to be present, encompassing organizational, technical, and practical aspects.

Consequently, the Hypno-TEC study aims to assess the feasibility of using virtual reality hypnosis (VRH) headset for anxiolytic purposes during frozen embryo transfer (FET).

Hypno-TEC will be a prospective interventional study, not comparative, and conducted at a single center, within the Reproductive Medicine Department of the Mother-Child-Woman Hospital in Lyon. This clinical investigation will fall under category 4.2 of medical device regulations, according to European Regulation 2017/745.

The enrolled patients, estimated to be 50 in number, will benefit from the device (VRH headset) during the execution of the FET procedure.

Besides assessing the feasibility of this usage, secondary outcomes will include: (i) evaluating the procedure's acceptability, (ii) patient and caregiver satisfaction with this application, (iii) effect on patient anxiety, and (iv) the pregnancy rates following the transfers concerned by the study.

The expected benefit is the potential to incorporate these headsets into routine practice, thereby would be enhancing patient adherence and tolerance to the transfer procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female patient aged between 18 and 45
* Currently undergoing In Vitro Fertilization treatment at the Assisted Reproduction Unit of the Mother-Child-Woman Hospital in Lyon
* Having a frozen embryo transfer planned, and for which the companion plans to be present
* Having signed an informed consent form
* Affiliated with the French social security system
* Understanding the French language, both spoken and written

Exclusion Criteria:

* Unbalanced epilepsy
* Patients with psychiatric disorders documented in their medical records
* Visual impairments preventing use of virtual reality (lack of binocular vision)
* Hearing impairments preventing use of audio headset (deafness, blindness)
* Claustrophobia
* First embryo transfer
* Fresh embryo transfer
* Persons under guardianship, curatorship or judicial protection
* Individuals deprived of liberty, persons receiving psychiatric care, and individuals admitted to a health or social facility for purposes other than clinical investigation
* Any medical condition judged by the investigator's expertise as incompatible with the research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
The feasibility of using a virtual reality hypnosis headset for anxiolysis during a frozen embryo transfer | The composite criterion will be assessed through three binary questions (corresponding to the three constituent criteria) to be answered by the FET operator immediately after the procedure.
  This is a combined criterion, requiring the validation of the following three criteria for the utilization of these headsets to be considered "feasible":
  * Availability of the headset on the day of the FET (yes/no)
  * Provision of the headset by the caregiver of the FET (yes/no)
  * Optimal use of the headset during the FET (yes/no) (i.e., optimal use is defined as the absence of technical incidents or battery depletion throughout the headset's usage duration during the procedure) A negative response to any of these three criteria will result in the procedure being deemed not feasible

SECONDARY OUTCOMES:
Duration of medical device usage (number of minutes) | This information will be collected by the FET operator immediately after FET.
  The duration will be estimated by the difference between the time of setting up the medical device and the time of removing the headset.
Measurement of procedure acceptability from the patients' perspective | This information will be completed by the patient immediately after the FET.
  It will be determined by the presence or absence of adverse effects experienced during the use of the device, collected through a binary question to which the patient will respond.
  In case of a positive response, the adverse effects will then be described, based on a (non-exhaustive) list provided to the patient, along with a declarative item if the adverse effect is not present in the list.
Satisfaction rate of patient regarding the procedure. | This information will be completed by the patient immediately after the FET.
  The assessment of satisfaction related to the use of the VRH headset will be measured using a Likert scale (very satisfied/satisfied/no opinion/dissatisfied/very dissatisfied).
Satisfaction rate of healthcare providers regarding the procedure. | This information will be completed by the caregiver immediately after the FET.
  The assessment of satisfaction related to the use of the VRH headset will be measured using a Likert scale (very satisfied/satisfied/no opinion/dissatisfied/very dissatisfied).
Effect of VRH headset usage on patient anxiety, measured through the change in average anxiety score | The 〖"STAI-Y1" 〗_"STATE " self-assessment anxiety questionnaire will be provided to the patient in paper format just before the FET and immediately after the procedure.
  Comparison of the average anxiety score measured using the 〖"STAI-Y1" 〗_"STATE " , before and after device usage.
Rate of biological pregnancies obtained after the FETs | This information will be obtained by reviewing the electronic medical records of the patients 1 month after the FET.
  The proportion of patients who have achieved a biological pregnancy will be determined by collecting the systematically performed HCG level measurement 10 days after the transfer.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No